CLINICAL TRIAL: NCT07062718
Title: Effects of Median Nerve Flossing Technique on Pain,Range of Motion and Disability in Patients With Cervical Radiculopathy
Brief Title: Median Nerve Flossing Technique in Patients With Cervical Radiculopathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0169
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Cervical Radiculopathy
Keywords: pain; range of motion; disability
MeSH Terms: conditions — Radiculopathy; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Median nerve flossing technique and conventional physical therapy (Active Comparator): Nerve flossing will be started from root along brachial plexus,median nerve root.
  Before starting the procedure ,subjects will be shown the flossing technique as it will be performed actively by the subjects. Each flossing will be performed with 10 repetitions starting from neck,arm,elbow,wrist and whole nerve flossing (12).
  It will be a 3 week treatment with 4 session per week (12 sessions) (12).
  Interventions: Other: Median nerve flossing technique and conventional physical therapy
- Conventional physical therapy (Active Comparator): The subjects in this group will be treated with TENS and hot pack. All the subjects will be screened according to the inclusion and exclusion criteria .Written informed consent will be taken from all the subjects before the treatment. The subjects will be allowed to withdraw the treatment any time.The subjects will be divided into 2 groups through convenience sampling.All the subjects from both group will be given trancutaneous electric nerve stimulation TENS ,hot pack, isometrics and stretching as a conventional physical therapy followed by respective group techniques
  The session will last for 20 -25 minutes , TENS pad will be placed in the suboccipital region and the trapezius unilaterally with hot pack simultaneously for 10 minutes
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Median nerve flossing technique and conventional physical therapy — Median nerve flossing technique and conventional physical therapy Nerve flossing will be started from root along brachial plexus,median nerve root.
  Before starting the procedure ,subjects will be shown the flossing technique as it will be performed actively by the subjects. Each flossing will be performed with 10 repetitions starting from neck,arm,elbow,wrist and whole nerve flossing (12).
  It will be a 3 week treatment with 4 session per week (12 sessions)
  Other Names: conventional physical therapy
  Arms: Median nerve flossing technique and conventional physical therapy
Other: Conventional physical therapy — The subjects in this group will be treated with TENS and hot pack. All the subjects will be screened according to the inclusion and exclusion criteria .Written informed consent will be taken from all the subjects before the treatment. The subjects will be allowed to withdraw the treatment any time.The subjects will be divided into 2 groups through convenience sampling.All the subjects from both group will be given trancutaneous electric nerve stimulation TENS ,hot pack, isometrics and stretching as a conventional physical therapy followed by respective group techniques
  The session will last for 20 -25 minutes , TENS pad will be placed in the suboccipital region and the trapezius unilaterally with hot pack simultaneously for 10 minutes
  Arms: Conventional physical therapy

SUMMARY:
Cervical radiculopathy is a condition of cervical spinal nerve roots which occurs as a result of compression and inflammatory pathology from a space occupying lesion. Nerve flossing technique is a quick mobilization of the strained nerves which will reduce pain .This study aim to determine the effects of nerve flossing technique on pain, range of motion and disability in patients with cervical radiculopathy.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial and will be conducted in Riphah Rehabilitation Clinic Lahore and Shalamar Hospital(physiotherapy department) Lahore. Non-probability convenient sampling will be used to collect the data. Sample size of 38 subjects with age group between 30 to 50 years will be taken. Data will be collected from the patients having unilateral median nerve symptoms of cervical radiculopathy. Outcome measures will be taken using Numeric pain rating scale(NPRS) for pain, Neck disability index (NDI) and Universal Goniometer (GU) for Range of motion. An informed consent will be taken. Subjects will be selected on the basis of inclusion and exclusion criteria and will be equally divided into two group by convenience sampling. Both the Groups will receive Transcutaneous electrical nerve stimulation (TENS), Hot Pack, cervical isometric and cervical stretching , while Group A will receive conventional treatment and Group B will receive an additional nerve flossing technique. Outcome measures, Numeric Pain Rating scale (NPRS) for pain ,Neck Disability Index (NDI) for disability and Universal Goniometer for range of motion will be measured at baseline and after 3 weeks of treatment total 12 sessions(4 sessions per week ).Data analysis will be done by SPSS version 21.0.

ELIGIBILITY:
Inclusion Criteria:• Both male and female gender were included

* Participants with 30 to 50 years of age group were taken in this study (Gore et al., 2020)
* Patients with positive Spurling test ,cervical distraction ,cervical rotation test were included
* Participants with positive Upper limb neural tension test for median nerve were taken into consideration
* Patients who are having radicular symptoms and pain for more than 3 months were included

Exclusion Criteria:

* Systematic disorders affecting musculoskeletal disorders e.g. Ankylosing spondylitis,rheumatic arthritis etc.
* Patient with primary shoulder or upper limb pain origin
* Patients with severe malignancy,COPD ,isch

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-07-25 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
numeric pain rating scale | 4 weeks
  The intensity of pain was assessed with the help of NPRS. The scale have readings that numerate from 0 to 10,beginning with least reading 0 that indicates no pain ,5 indicates moderate level of pain and 10 indicates extreme level of pain.Test-retest reliability of NPRS was high

SECONDARY OUTCOMES:
goniometer | 4 weeks
  Universal goniometer was used to measure range of motion of cervical region that has an inter-rater reliability

OTHER OUTCOMES:
universal goniometer | 4 weeks
  Disability level of neck was demonstrated by using Neck Disability Index (NDI) questionnaire .It consist of total 10 sections, each with 0-5 rating scale in which 0 indicates "

CONTACTS AND LOCATIONS:
Overall Officials: Asif Sheikh, MBBS FCPS, Study Chair — Pediatric clinic
Locations (1):
- Dr Asif Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anandkumar S. The effect of sustained natural apophyseal glide (SNAG) combined with neurodynamics in the management of a patient with cervical radiculopathy: a case report. Physiother Theory Pract. 2015 Feb;31(2):140-5. doi: 10.3109/09593985.2014.971922. Epub 2014 Oct 20. PMID 25329587
- [Background] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561
- [Background] Cleland JA, Childs JD, McRae M, Palmer JA, Stowell T. Immediate effects of thoracic manipulation in patients with neck pain: a randomized clinical trial. Man Ther. 2005 May;10(2):127-35. doi: 10.1016/j.math.2004.08.005. PMID 15922233
- [Background] Dimitrov, T., Hussain, N., & Abd-Elsayed, A. (2022). Median Nerve. Peripheral Nerve Stimulation-E-Book: A Comprehensive Guide, 82.
- [Background] Farooq MN, Mohseni Bandpei MA, Ali M, Khan GA. Reliability of the universal goniometer for assessing active cervical range of motion in asymptomatic healthy persons. Pak J Med Sci. 2016 Mar-Apr;32(2):457-61. doi: 10.12669/pjms.322.8747. PMID 27182261
- [Background] Gore, V., Patil, H., & Chogule, A. (2020). Effect of Cervical Manual Traction, TENS and Neural Tissue Mobilization on Pain and Functional Disability in Unilateral Cervical Radiculopathy. Website: Www. Ijrrjournal. Com Original Research Article International Journal of Research and Review (Ijrrjournal. Com), 7(10), 198-200.
- [Background] omparison of Treatment Outcome of the Effectiveness of Isometric Exercises as Hayat, M., Siddique, R., Basharat, A., Waheed, I., Rubab, S. U., Naqvi, H., . . . Haq, F. (2023). Compared to General Exercises with Cervical Spine Mobilization in The Management of Chronic Non Specific Neck Pain. British Journal of Multidisciplinary and Advanced Studies, 4(6), 63-72.
- [Background] Kage, V., & Gurav, G. (2017). Effect of neural flossing technique on pain, cervical range of motion and functional ability in subjects with acute, sub-acute trapezitis: An experimental study. Int. J. Appl. Res, 3, 818-822.
- [Background] Karkousha, R. N., Selem, A. I., Aly, S. A., & Zahran, M. R. (2023). Mulligan mobilization technique versus neural mobilization on nerve root function in patients with cervical radiculopathy: Randomized controlled trial. Revista iberoamericana de psicología del ejercicio y el deporte, 18(6), 670-675.